CLINICAL TRIAL: NCT05920070
Title: Therapeutic Mammoplasty Doesn't Delay Adjuvant Therapy for Breast Cancer Patients
Brief Title: the Effect of Therapeutic Mammoplasty on the Start of Adjuvant Chemotherapy
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Nabil Anwer, resident at general surgery department, Assiut University
Other Study IDs: tmp and adjuvant chemotherapy
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Effect of Therapeutic Mammoplasty on Adjuvant Chemotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: therapeutic mammoplasty — therapeutic oncoplastic surgeries in cases of breast cancer

SUMMARY:
the purpose of this study was to examine the impact of therapeutic mammoplasty on the delivery of adjuvant chemotherapy

DETAILED DESCRIPTION:
One out of every eight women will be diagnosed with breast cancer in her lifetime, making it the most common cancer in women. Over the last decades the survival rate has increased slowly, which is currently estimated to be 85 % in developed countries. However, with an estimated annual number of breast cancer deaths of 537,000 worldwide, breast cancer still is the most important cause of death by cancer among women. Despite advances in different treatment modalities, about 45 % of all breast cancer patients still undergoes a mastectomy for adequate local control. The resulting loss of a breast may have a negative effect on body image, sexuality, and sense of femininity. (8) Oncoplastic breast techniques are being increasingly employed to allow breast conservation whilst maintaining a quality aesthetic outcome. Therapeutic mammoplasty (TM) describes multiple breast-conserving techniques1 which remove the breast tumour in combination with adjuvant radiotherapy (1). TM is available to women with early stage breast cancer with larger or ptotic breasts who would benefit from a reduction mammoplasty technique in addition to tumour removal. The use of TM is increasing worldwide, with the potential to deliver benefits both oncologically, in terms of increased tumour free margin width, and with an associated superior long-term aesthetic outcome. Despite increasing enthusiasm for the techniques there is limited data on long-term oncological safety or effects upon delivery of adjuvant treatments.TM techniques can enable a larger volume of tissue to be resected with the tumour6 enabling patients to have breast-conserving surgery for larger tumours. Just as the role of TM is expanding, adjuvant chemotherapy is increasingly being used in women with early stage breast cancer and if delivered in a timely fashion after the primary resection, decreases recurrence and improves overall survival (3). However, TM is associated with higher complication rates than traditional breast-conserving methods and one barrier to TM is the concern that post-operative complications may lead to a delay in initiation of chemotherapy or even omission. There is increasing evidence that immediate breast reconstruction has an effect on adjuvant chemotherapy delivery. Three recent series involving over 4000 patients suggest that immediate breast reconstruction does lead to a significant delay in the delivery of adjuvant chemotherapy (2). However, the clinical significance of this delay has not been established. On the contrary, a recent study performed by Doughty et al. compared 95 patients undergoing immediate breast reconstruction following mastectomy with cohorts having breast-conserving surgery and simple mastectomy with no reconstruction, in which no delay to commencement of adjuvant chemotherapy was noted. The majority of case series on TM do not comment on the timing of adjuvant treatments. When they are reported, studies vary between no delays to adjuvant treatment through to five studies reporting delays in between 1.9%9 and 6% of patients (8).

ELIGIBILITY:
Inclusion Criteria:

* Oncoplastic procedures were proposed for patients in whom breast conservative treatment is possible on oncologic grounds but in whose cases a standard resection without reconstruction would result in poor cosmesis with the following criteria:

  1. Female patients with ages ranging from 25 to 65 years
  2. Patients with early surgically treatable breast cancer (Stage I, II and IIIa)
  3. Patients whose management was by surgery followed by adjuvant chemotherapy.
  4. Patients with tumors in any quadrant of the breast
  5. Patients with large/ptotic breasts (especially with brassiere size C, D or DD).
  6. patients underwent therapeutic mammoplasty as primary ttt for breast cancer.

Exclusion Criteria:

* 1) Patients with a contraindication to breast conservative surgery. 2) Patients with small sized breasts, which are not suitable for reduction (with brassiere size A or B).

  3) Patients who are not compliant; Non-compliant patients included those demanding mastectomy for fear of local recurrence, patients not consenting to the proposed procedure after adequate counseling, those refusing post-operative adjuvant Radiotherapy, refusal of a reduction mammoplasty of the contralateral breast as a symmetrizing procedure and patients who are not able to consent such as mentally challenged patients.

  4) patients who have received neoadjuvant chemotherapy. 5) patients underwent conventional breast conservative surgery . 6) patient underwent immediate reconstruction surgery.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female patient underwent therapeutic mammoplasty
Study Population: female patients between the age of 25 to 65 who underwent therapeutic ammoplasty and will recieve adjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
assesing the complocation of therapeutic mammoplasty and whether it delays the start of adjuvant chemotherapy or not | about two months
  noting the date of the operation and whether or not it delays the start of adjuvant chemotherapy due to any complications

CONTACTS AND LOCATIONS:
Overall Officials: abdelradi amdelsalam, proffessor, Study Director — Assiut University; mostapha thabet, professor, Study Director — Assiut University; negmeldeen abulnaga, assistant lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: about two years

REFERENCES:
- [Result] Harvey J, Henderson J, Patel L, Murphy J, Johnson R. Therapeutic mammaplasty - impact on the delivery of chemotherapy. Int J Surg. 2014;12(5):51-5. doi: 10.1016/j.ijsu.2013.10.013. Epub 2013 Nov 5. PMID 24200754
- [Result] Bamford R, Sutton R, McIntosh J. Therapeutic mammoplasty allows for clear surgical margins in large and multifocal tumours without delaying adjuvant therapy. Breast. 2015 Apr;24(2):171-4. doi: 10.1016/j.breast.2015.01.003. Epub 2015 Jan 24. PMID 25623754
- [Result] Khan J, Barrett S, Forte C, Stallard S, Weiler-Mithoff E, Doughty JC, Romics L Jr. Oncoplastic breast conservation does not lead to a delay in the commencement of adjuvant chemotherapy in breast cancer patients. Eur J Surg Oncol. 2013 Aug;39(8):887-91. doi: 10.1016/j.ejso.2013.05.005. Epub 2013 Jun 5. PMID 23746877
- [Result] 4. Simpson, Gregory, M. Chandrashekar, and S. Darn.
- [Result] Dogan L, Gulcelik MA, Karaman N, Ozaslan C, Reis E. Oncoplastic surgery in surgical treatment of breast cancer: is the timing of adjuvant treatment affected? Clin Breast Cancer. 2013 Jun;13(3):202-5. doi: 10.1016/j.clbc.2012.09.015. Epub 2012 Oct 26. PMID 23103367
- [Result] Klit A, Tvedskov TF, Kroman N, Elberg JJ, Ejlertsen B, Henriksen TF. Oncoplastic breast surgery does not delay the onset of adjuvant chemotherapy: a population-based study. Acta Oncol. 2017 May;56(5):719-723. doi: 10.1080/0284186X.2017.1281437. Epub 2017 Feb 6. PMID 28162018
- [Result] Kontos M, Lewis RS, Luchtenborg M, Holmberg L, Hamed H. Does immediate breast reconstruction using free flaps lead to delay in the administration of adjuvant chemotherapy for breast cancer? Eur J Surg Oncol. 2010 Aug;36(8):745-9. doi: 10.1016/j.ejso.2010.06.013. PMID 20605080